CLINICAL TRIAL: NCT02564822
Title: Effects of the Visual Stimulation on the Motor and Visual Cortex in Migraneurs With and Without Aura
Status: Completed | Type: Observational
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, Kátia Monte-Silva, Principal Investigator, Universidade Federal de Pernambuco
Other Study IDs: VisualStimulation_Migraine
Record Dates: First submitted 2015-09-22; First posted 2015-10-01 (Estimated); Last update posted 2018-08-24 (Actual); Status verified 2018-08

CONDITIONS: Migraine Disorders
Keywords: migraine disorders; cortical excitability; transcranial magnetic stimulation; electroencephalography
MeSH Terms: conditions — Migraine Disorders | interventions — Photic Stimulation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Migraneurs - Visual stimulation: Patients will be recruited via advertisements on the university. Patients should have migraine diagnosis according to the International Classification of Headache Disorders (ICHD-III) criteria and clinical diagnosis by a neurologist.
  Interventions: Procedure: Visual Stimulation
- Control - Visual stimulation: Healthy volunteers will be recruited via advertisements on the university. For control subjects the individuals should not have migraine diagnosis assessed according to IHCD-III criteria.
  Interventions: Procedure: Visual Stimulation

INTERVENTIONS:
Procedure: Visual Stimulation — volunteers will be invited to sit in a comfortable chair, in a calm and dark room, at 90 cm of distance from computer screen. It will be asked to fix his right eye visual field on a red point at the center of the screen (the left one will be blindfolded). Visual stimuli will be a black and White grid pattern, alternating at a frequency of 3.1 Hz.

SUMMARY:
The aim of this study is to investigate the motor and visual cortex excitability in response to visual stimulation of migraineurs with and without aura compared to healthy individuals. For this purpose, electrical cortical activity of migraineurs will be compared to healthy volunteers.

DETAILED DESCRIPTION:
A cross sectional study to compare the best approach to migraineurs evaluation. For this, healthy individuals, after reading and signing the free and informed consent will be submitted to a single session to obtain the normal neurophysiological endpoints and thus compare with those obtained in individuals with migraineurs volunteers. All volunteers (healthy and migraineurs) will be submitted to a neurophysiological evaluation through transcranial magnetic stimulation (TMS) and electroencephalography (EEG). A visual stimulation will be delivered during the assessment of habituation through visual evoked potential volunteers (VEP-habituation) and the following measures will be evaluated before and after visual stimulation: (i) Motor Evoked Potentials (MEP); (ii) Motor Threshold (MT); (iii) Short Interval Cortical Inhibition (SICI); (iv) Intracortical Facilitation (lCF) and (v) Phosphene Threshold (PT).

ELIGIBILITY:
Inclusion Criteria:

* Ages: 18-55 years
* Gender: Both
* Prior headache report

Exclusion Criteria:

* Pregnant women;
* Pacemaker;
* History of seizures;
* Metallic implants in the head;
* Patients with clinical evidence of brain injuries;
* Chronic pain associated to others diseases;
* Use of neuroleptic medications

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients and healthy volunteers will be recruited via advertisements on the university. Patients should have migraine diagnosis according to the International Classification of Headache Disorders (ICHD-III) criteria and clinical diagnosis by a neurologist.
  For control subjects the individuals should not have migraine diagnosis assessed according to IHCD-III criteria.
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Changes on motor evoked potentials | one day (Before and after visual stimulation)
  to measure MEP, the intensity of the magnetic stimulator will be adjusted to 120% of rest motor threshold and 10 stimuli will be registered. For evaluation volunteers will be instructed to sit in a chair and get into a comfortable position. Initially, single-pulse TMS will be administered over the motor cortex to determine the cortical representation area of the first dorsal interosseous muscle (FDI). For all evaluations the same figure-eight coil is used, in order to avoid measurement bias. Amplitude means of evoked potentials will determine the MEP.

SECONDARY OUTCOMES:
Changes on short interval intracortical inhibition | one day (Before and after visual stimulation)
  to evaluate this variable, subthreshold conditioning stimuli (80% of RMT) and suprathreshold test stimuli (120% of RMT) will be delivered at an inter stimulus intervals (ISI) of 2 milliseconds, to determine the short interval cortical inhibition (SICI). Ten stimuli will be applied in each condition (unconditioned pulse and pairs of stimuli with ISI of 2 milliseconds). The order of stimulus delivered will be pseudorandomized and SICI will be expressed as a percentage of a conditioned stimuli in regarding an unconditioned stimuli.
Changes on intracortical facilitation | one day (Before and after visual stimulation)
  to evaluate intracortical facilitation (ICF), subthreshold conditioning stimuli (80% of RMT) and suprathreshold test stimuli (120% of RMT) will be delivered at an inter stimulus intervals (ISI) of 10 milliseconds. Ten stimulus will be applied in each condition (unconditioned pulse and pairs of stimuli with ISI of 10 milliseconds). The order of stimuli delivered will be pseudorandomized and ICF will be expressed as a percentage of a conditioned stimuli in regarding an unconditioned stimuli.
Changes from phosphene threshold | one day (Before and after visual stimulation)
  a 10-cm circular coil was used that has giving a peak magnetic field strength of 2 tesla. Subjects were asked to wear a blindfold, sit comfortably in a chair and to close their eyes to diminish ambient light.In sagittal line, three points were scored: 2, 3 and 4 cm above the inion. The single pulse TMS was applied to one of the points scored and the subject was asked to report the presence or absence of a phosphene immediately after stimulation. The stimulation was repeated ten times at each intensity with a maximum frequency of 0.2 Hz, stimulation was initially applied to 60% of the maximum intensity of the stimulator. The intensity of stimulation was changed into blocks of 5% to minimum intensity that the subject can perceive the phosphene certainly, five times ten, then this value was set as the PT.
Habituation of Visual Evoked Potentials evaluated by Electroencephalography | one day (during visual stimulation)
  volunteers will be invited to sit in a comfortable chair, in a calm and dark room, at 90 cm of distance from computer screen. It will be asked to fix his right eye visual field on a red point at the center of the screen (the left one will be blindfolded). Visual stimuli will be a black and White grid pattern, alternating at a frequency of 3.1 Hz. Electrodes used to record data will be localized on Oz and Fz points according International 10-20 system. During the test, 600 cortical answers will be recorded. Data will be collected and recorded in a personal computer, and after, converted to the ".txt" format to futures analysis with MATLAB.

CONTACTS AND LOCATIONS:
Overall Officials: Kátia Monte-Silva, PhD, Principal Investigator — Universidade Federal de Pernambuco
Locations (1):
- Laboratório de Neurociência Aplicada (LANA), Recife, Pernambuco, Brazil